CLINICAL TRIAL: NCT06359392
Title: Culturally Responsive Palliative Care Messaging for American Indians: An Efficacy Trial
Brief Title: Palliative Care Messaging for American Indians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Collaborators: Great Plains Tribal Leaders Health Board (Unknown); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mary Isaacson, Associate Professor, South Dakota State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DNZNC466DGR7; 1R21NR020383-01 (NIH)
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: palliative care; American Indian; hospice; end of life
MeSH Terms: conditions — Behavior; Death | interventions — NMT1 protein, S pombe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Message (Other): Individuals assigned to this arm will take the surveys only and not be exposed to a palliative care message.
  Interventions: Other: No message
- Culture-centric message (Other): Individuals assigned to this arm will watch a 2 minute culture-centric palliative care video specific for these American Indian communities and then take the surveys after watching the videos.
  Interventions: Other: Culture-centric message
- General message (Other): Individuals assigned to this arm will watch a 2 minute palliative care video created for the general US population and then take the surveys after watching the videos.
  Interventions: Other: General messge

INTERVENTIONS:
Other: No message — Participants will not be exposed to a message in this arm of the intervention.
  Arms: No Message
Other: Culture-centric message — Participants in this arm of the study will watch a 2-minute video on palliative care developed specifically for these American Indian communities.
  Arms: Culture-centric message
Other: General messge — Participants receiving this intervention will watch a 2-minute video developed by the National Hospice and Palliative Care Organization to teach about palliative care.
  Arms: General message

SUMMARY:
The investigators will be conducting a randomized trial in 3 reservation communities to test the efficacy of the narrative as culture-centric health promotion model for increasing American Indian tribal members' palliative care knowledge and intentions to discuss palliative care.

DETAILED DESCRIPTION:
Palliative care is specialized patient-/family-centered care designed to reduce suffering and enhance quality of life for persons with serious illness. Culturally responsive palliative care can ease serious illness burden experienced by American Indians (AIs) and improve seriously ill AIs end-of-life decision-making. However, for seriously ill Northern Plains AIs, specifically those in South Dakota (SD), access to and use of culturally responsive palliative care is severely limited. To address this need, the investigators have formed a multidisciplinary, tribally-driven collaborative team consisting of Great Plains Tribal Leaders Health Board, active AI community advisory boards at the following reservations: Cheyenne River, Rosebud, and Pine Ridge, and South Dakota State University. The research team will conduct a campaign messaging efficacy test using the narrative as culture-centric health promotion model (NCHP) to create and test culture-centric narrative messaging that improves knowledge of palliative care and encourages participants to engage in formal and informal communication about palliative care. The NCHP model is an evidence-based innovative approach to enhance AI's knowledge and intentions to talk formally and informally about palliative care, because it provides guidelines for how to construct culture-centric narratives which identify the features of effective narratives and the mechanisms by which the narratives work to transform cognitive and behavioral outcomes. The investigators have developed a culture-centric narrative health video message and will be conducting a randomized trial to test the efficacy of the NCHP model for increasing AI tribal members' palliative care knowledge and intentions to discuss palliative care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Self-identify as American Indian
* Must be able to read and comprehend English
* Live on or around the Pine Ridge Indian Reservation, Rosebud Indian Reservation, or Cheyenne River Indian Reservation

Exclusion Criteria:

* Under the age of 18 years
* Not American Indian
* Do not live near or on the Pine Ridge Indian Reservation, Rosebud Indian Reservation, or Cheyenne River Indian Reservation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Palliative Care Knowledge Scale (PaCKS) | 2 hours
  The 13-item PaCKS measures palliative care knowledge among lay people, using true/false items covering topics like goals of palliative care. We know palliative care awareness is lacking; thus it is important to understand knowledge gaps; hence we will modify the response options to include "I don't know" in addition to true/false.
Knowledge of Care Options (KOCO) | 2 hours
  The 11-item KOCO measures gaps in knowledge of care options among cancer patients for curative, palliative, and hospice care using true-false options.
Hospice and Palliative Care Questionnaire (HPCQ) | 2 hours
  The 12-item HPCQ examines attitudes, use, and interest in receiving more information. There are 6 hospice and 6 palliative care questions, that have been used successfully with ethnically diverse populations.
Identification and Transportation with Palliative Care Message | 2 hours
  Individuals watching either the culture-centric palliative care video or the general video will be asked to ask 5 questions about emotions they felt, how they identified with the main characters in the video, and how focused they were while watching the video
Attitudes and Intentions to Discuss Palliative Care | 2 hours
  Those watching the culture-centric video or the general message video will be asked to respond to 5 questions about their intentions to discuss pallative care with their family.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Isaacson, PhD, RN, Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Rapid City, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
We are working with Tribal communities that are sovereign nations and we will share their data back with them at the end of the trial. We have to obtain special permission in order to share de-identified data more broadly.